CLINICAL TRIAL: NCT01403428
Title: Effect Of Early Initiation Of Noninvasive Positive Pressure Ventilation On ICU Length Of Stay In Children With Status Asthmaticus, A Prospective Randomized Trial
Brief Title: Non Invasive Positive Pressure Ventilation in Status Asthmaticus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In a pilot of early noninvasive positive pressure ventilation, the children did so well that early NPPV is now used in all children who meet criteria.
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAS-SIU-11-005
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Status Asthmaticus
Keywords: Asthma; non invasive ventilation; pediatrics; noninvasive positive pressure ventilation (NPPV)
MeSH Terms: conditions — Status Asthmaticus; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPPV plus standard of care (Experimental): Noninvasive positive pressure ventilation (NPPV) plus standard of care in the management of children admitted to the hospital with status asthmaticus
  Interventions: Other: Noninvasive positive pressure ventilation
- Standard of care (No Intervention): standard of care treatment in the management of children admitted to the hospital with status asthmaticus

INTERVENTIONS:
Other: Noninvasive positive pressure ventilation — Noninvasive positive pressure ventilation (NPPV) will deliver pressurized gas through a nasal or oronasal mask, connected to a pressure targeted ventilator. NPPV provides ventilator support without the use of an endotracheal tube. Standard of care includes use of corticosteroids, oxygen, short acting β-agonist and inhaled ipratropium bromide.
  Arms: NPPV plus standard of care

SUMMARY:
Status Asthmaticus is recognized as a common cause of morbidity in children in the United States (CDC). In recent years, hospitalization rates have reached an all time high. This study will evaluate the effect of early use of noninvasive positive pressure ventilation (NPPV) in children admitted to the pediatric intensive care unit (PICU) with moderate to moderately severe status asthmaticus to test the hypothesis that early initiation of NPPV plus standard of care will result in decreased length of PICU stay, significant improvement in clinical asthma score (CAS) and reduced patient care costs when compared to standard of care alone.

DETAILED DESCRIPTION:
Asthma is a common, chronic and complex disorder of the airways, with symptoms that are variable and recurring. It is characterized by bronchial hyper-responsiveness to various stimuli, airflow obstruction that is often reversible, and underlying inflammation. Conventional therapy for status asthmaticus is directed at relieving broncho-constriction, decreasing airway inflammation and clearing airway mucus. However, in some patients, maximal standard therapies are inadequate and can lead to prolonged hospitalization. Intubation and mechanical ventilation in patients with asthma is associated with significant risks. NPPV has several advantages over invasive intubation and mechanical ventilation. It leaves the upper airway intact, and avoids the risks associated with endotracheal intubation including upper airway trauma, laryngeal swelling, postextubation vocal cord dysfunction, and nosocomial infections.

This study will be a prospective, open-labeled, randomized clinical trial comparing the use of NPPV plus standard of care versus standard of care alone in children admitted for status asthmaticus. A simple random numbers table will be used to assign subjects to either the NPPV plus standard of care group or standard of care alone group. In the first hour, all patients in both groups will receive a 2mg/kg dose of systemic steroid, continuous albuterol at 0.5mg/kg/hr (max of 15mg/hr) with 3 doses of 0.25-0.5 mg nebulized ipratropium bromide, and supplemental oxygen keep saturation >92%. Patients on both therapeutic arms will continue to receive 2mg/kg dose of systemic steroid per day, continuous albuterol at 0.5mg/kg/hr (max of 15mg/hr) and supplemental oxygen to keep saturation >92%.

Patients randomized to the NPPV plus standard of care group will be fitted with a nasal or face mask and placed on the Respironics V60 bilevel positive airway pressure (BiPAP) Ventilator 33. Masks with gel seals at different pressure points will be used to prevent skin breakdown. To optimize patient cooperation, the mask will initially be applied manually to the patient's face. After a short adaptation period for the patient to feel comfortable, the mask will be firmly applied with head straps to minimize air leak without causing skin injury. Pressures will initially be low for comfort and acceptance while being placed on the machine.

Patients randomized to the standard of care group will be placed on a similar continuous nebulizer attached to a similar oxygen blender as the ones used with the V60 unit set-up, using the same liter flow (11 liters per minute). An aerosol mask will be placed on the patient to aid in the delivery of the medication. The oxygen will be analyzed at the site of this mask with the initial set-up and any time the oxygen is decreased or increased.

Data will be collected at baseline as soon as the patient is enrolled in the study. It will include: demographic variables, medical record number, age, race, gender; history and physical findings, other medical conditions, vital signs, oxygen saturation at baseline, CAS, peak flow in children >6 years of age, asthma severity prior to admission, NPPV settings, length of stay in the PICU, side effect profiles (tremor, tachycardia, agitation, nausea, nasal bridge pain, skin irritation/ulceration, gastric distension, dry eyes/mucosal dryness, sinus/ear pain, aspiration pneumonia, hypotension and pneumothorax).

Each child's participation in the study will end when the child is transferred from the PICU.

ELIGIBILITY:
Inclusion Criteria:

* 1-18 years old
* Known H/O asthma
* With status asthmaticus
* CAS score 2-8 after one dose of systemic steroid, 1 hour of continuous albuterol and 3 doses of ipratropium bromide.

Exclusion Criteria:

* No previous history of asthma.
* Absence of airway protective reflexes.
* Absence of respiratory drive.
* Problems with clearing oral secretions.
* Need for emergent intubation as determined by the attending physician.
* Facial or airway anomaly or injury precluding the use of tight fitting mask.
* Discretion of the attending physician depending on the severity of illness

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
length of stay | baseline until transfer from PICU
  Number of hours patient hospitalized in PICU

SECONDARY OUTCOMES:
clinical asthma score | baseline until transfer from PICU
  Clinical asthma score (CAS) will be recorded in 2 hour segments by clinical evaluation of 5 items-respiratory rate, inspiratory-expiratory ratio, retractions, adequacy of air exchange and wheezing-on a 3-point scale. A higher score indicates worsening respiratory status.
tolerability | baseline until transfer from PICU
  Number of hours patient able to wear the NPPV mask will be recorded in 2 hour segments.
patient care costs | baseline until transfer from PICU
  Actual costs accrued during PICU stay.
safety | baseline until transfer from PICU
  measure of clinical monitoring parameters:
  * Respiratory rate
  * pH
  * PaCO2

CONTACTS AND LOCATIONS:
Overall Officials: Sangita Basnet, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States

REFERENCES:
- See also: Southern Illinois University School of Medicine website — http://www.siumed.edu/
- See also: St. John's Children's Hospital — http://www.st-johns.org/childrensHospital/main/default.asp
- See also: American Lung Association - asthma webpage — http://www.lungusa.org/lung-disease/asthma/